CLINICAL TRIAL: NCT03045731
Title: An US Mathematical Model in Predicting Renal Transplant Rejection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FDU-ZS-US-001
Record Dates: First submitted 2017-01-14; First posted 2017-02-07 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; ultrasound; mathematical model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Kidney transplant recipients: Patients who have received kidney transplantation in Zhongshan Hospital.

SUMMARY:
The purpose of this study is to establish an ultrasound mathematical model using acoustic radiation force impulse (ARFI) and contrast-enhanced ultrasonography (CEUS) for diagnosing the status of renal allografts.

DETAILED DESCRIPTION:
* There are various reasons for renal failure after kidney transplantation, such as delayed graft function (DGF) and acute rejection, acute renal tubular necrosis, chronic rejection and toxicity of immunosuppressive drugs. The diagnosis of renal allografts dysfunction can determine the direction of therapy. Currently, the gold standard of diagnosing renal allografts status is biopsies. However, biopsy has several drawbacks. It is invasive and can cause serious complications. These drawbacks urge investigators to find an accurate and non-invasive method to detect renal function. Elastography is a new way to detect tissue elasticity and can evaluate the tissue elasticity quantitatively. This method is proved to be of great value in diagnosing hepatic fibrosis (≥stage 2). Even though the investigation about this method is relatively less in allograft, the recent research shows that tissue elasticity does have relationship with pathological changes of transplanted kidney. Another new method, contrast-enhanced ultrasonography (CEUS), can indicate the blood perfusion of organ microcirculation. The accuracy rate of diagnosis of acute rejection(AR) can be 80% by using this method. It also has advantage in diagnosing acute tubular necrosis(ATN) and CAN. In addition, it produces no radioactive contamination as well as renal toxicity. This method has no serious side effect so it will not influence the normal function of patients' bodies and it can be performed for many times easily.
* The research information about Elastography and CEUS is still at the primary stage. The value of one single parameter in diagnosing renal failure is restricted. So the establishment of an integrated mathematical model got by combining traditional methods (such as ultrasonography and color Doppler flow imaging) with these two new methods (Elastography and CEUS) is required to provide a systematical, multi-parameter diagnosis of allograft rejection.
* What investigators have investigated before shows that different pathological changes of renal allograft can lead to regular changes in shear wave speed (SWS) and hemodynamics. By in-depth study of these changes, investigators aim to develop a mathematical model to diagnose the status of renal allograft.
* To achieve this goal, the following things will be done:

  1. Investigators plan to enroll 100 renal transplant recipients .
  2. Before biopsy, these things will be done : a. Normal ultrasonography will be performed on transplanted kidney to measure their size, cortical thickness and vertebral body. b. Color Doppler flow imaging will be performed to see blood supply of transplanted kidney and resistive index (RI) of renal seg-mental will be measured. c. Contrast enhanced ultrasonography examination will be performed using Philips iU-22 ultrasonic apparatus with a C5-1 probe (Philips,Amsterdam, theNetherlands)with an intravenous bolus injection of 0.6-1.0mL SonoVue (Bracco, Milan, Italy). Area under curve (AUC), peak intensity (PI), time-to-peak (TTP), rise time (RT) and mean transit time (MTT) will be measured on central cortex of transplanted kidney. d. Elastography will be performed with a Siemens Acuson S2000 ultrasound machine using a 1- to 4-MHzcurved array multifrequency transducer (4 C1) (Siemens,Munich, Germany).

     Shear wave velocity (SWV) will be measured.
  3. Statistical analysis will be performed on the 10 quantitative parameters we got before (AUC, PI.etc ). The correlation between these parameters and condition of transplanted kidney (got by renal biopsy) will be evaluated. Then screening indexes will be optimized. On this basis, a mathematical model in diagnosing transplanted kidney is supposed to be built up.
  4. A ROC curve will be used to analyze the accuracy, sensitivity and specificity of this mathematical model.
  5. Then the US model will be verified in another 80 renal transplant recipients. Investigators will compare the diagnosis efficacy of transplanted kidney status got by the US model with the kidney biopsy result. Any parameter can be adjusted according to the verification results.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18) who have undergone renal transplant at Zhongshan Hospital
* Understanding the research situation
* Signing informed consent voluntarily

Exclusion Criteria:

* Urinary obstruction
* Perirenal hematioma
* Infection in operative sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (over 18) who have undergone renal transplant for at Zhongshan Hospital.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnosis of the status of kidney allografts from biopsy results | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Williams WW, Taheri D, Tolkoff-Rubin N, Colvin RB. Clinical role of the renal transplant biopsy. Nat Rev Nephrol. 2012 Jan 10;8(2):110-21. doi: 10.1038/nrneph.2011.213. PMID 22231130
- [Background] Schwenger V, Keller T, Hofmann N, Hoffmann O, Sommerer C, Nahm AM, Morath C, Zeier M, Krumme B. Color Doppler indices of renal allografts depend on vascular stiffness of the transplant recipients. Am J Transplant. 2006 Nov;6(11):2721-4. doi: 10.1111/j.1600-6143.2006.01524.x. PMID 17049059
- [Background] Hanamura K, Tojo A, Kinugasa S, Asaba K, Fujita T. The resistive index is a marker of renal function, pathology, prognosis, and responsiveness to steroid therapy in chronic kidney disease patients. Int J Nephrol. 2012;2012:139565. doi: 10.1155/2012/139565. Epub 2012 Dec 16. PMID 23304501
- [Background] Benozzi L, Cappelli G, Granito M, Davoli D, Favali D, Montecchi MG, Grossi A, Torricelli P, Albertazzi A. Contrast-enhanced sonography in early kidney graft dysfunction. Transplant Proc. 2009 May;41(4):1214-5. doi: 10.1016/j.transproceed.2009.03.029. PMID 19460520
- [Background] Grzelak P, Szymczyk K, Strzelczyk J, Kurnatowska I, Sapieha M, Nowicki M, Stefanczyk L. Perfusion of kidney graft pyramids and cortex in contrast-enhanced ultrasonography in the determination of the cause of delayed graft function. Ann Transplant. 2011 Jan-Mar;16(1):48-53. PMID 21436774
- [Background] Schwenger V, Korosoglou G, Hinkel UP, Morath C, Hansen A, Sommerer C, Dikow R, Hardt S, Schmidt J, Kucherer H, Katus HA, Zeier M. Real-time contrast-enhanced sonography of renal transplant recipients predicts chronic allograft nephropathy. Am J Transplant. 2006 Mar;6(3):609-15. doi: 10.1111/j.1600-6143.2005.01224.x. PMID 16468973
- [Background] Fierbinteanu-Braticevici C, Andronescu D, Usvat R, Cretoiu D, Baicus C, Marinoschi G. Acoustic radiation force imaging sonoelastography for noninvasive staging of liver fibrosis. World J Gastroenterol. 2009 Nov 28;15(44):5525-32. doi: 10.3748/wjg.15.5525. PMID 19938190
- [Background] Arndt R, Schmidt S, Loddenkemper C, Grunbaum M, Zidek W, van der Giet M, Westhoff TH. Noninvasive evaluation of renal allograft fibrosis by transient elastography--a pilot study. Transpl Int. 2010 Sep;23(9):871-7. doi: 10.1111/j.1432-2277.2010.01057.x. Epub 2010 Feb 15. PMID 20158692
- [Background] Stock KF, Klein BS, Vo Cong MT, Sarkar O, Romisch M, Regenbogen C, Buttner M, Schuster T, Matevossian E, Amann K, Clevert DA, Heemann U, Kuchle C. ARFI-based tissue elasticity quantification in comparison to histology for the diagnosis of renal transplant fibrosis. Clin Hemorheol Microcirc. 2010;46(2-3):139-48. doi: 10.3233/CH-2010-1340. PMID 21135489
- [Background] Fischer T, Filimonow S, Rudolph J, Morgera S, Budde K, Slowinski T, Ebeling V, Taymoorian K, Giessing M, Thomas A. Arrival time parametric imaging: a new ultrasound technique for quantifying perfusion of kidney grafts. Ultraschall Med. 2008 Aug;29(4):418-23. doi: 10.1055/s-2006-927269. Epub 2007 Feb 21. PMID 17315111
- [Background] Schwenger V, Zeier M. Contrast-enhanced sonography as early diagnostic tool of chronic allograft nephropathy. Nephrol Dial Transplant. 2006 Oct;21(10):2694-6. doi: 10.1093/ndt/gfl449. Epub 2006 Jul 28. No abstract available. PMID 16877483
- [Background] Scholbach T, Girelli E, Scholbach J. Dynamic tissue perfusion measurement: a novel tool in follow-up of renal transplants. Transplantation. 2005 Jun 27;79(12):1711-6. doi: 10.1097/01.tp.0000164145.89275.02. PMID 15973173